CLINICAL TRIAL: NCT03735303
Title: The Combined Effect of Vitamin D3 and Omega-3 Supplements on Serum Leptin and Glycated Hemoglobin (Hb A1C) Levels in Jordanian People With Vitamin D Deficiency.
Brief Title: Effect of Vitamin D3 and Omega-3FA on Leptin and HbA1C With Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DRGS-4-2018
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2018-12

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D3; vitamin D deficiency; leptin; A1C; omega-3 fatty acid
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VD3 group (Experimental): dietary supplement : VD3 group treated with 50000 IU VD3/ week for 8 weeks
  Interventions: Dietary Supplement: VD3 group
- omega 3- FA group (Experimental): dietary supplement : omega 3- FA group 1000 mg wild salmon and fish oil complex (contain 300 mg of omega 3-FA) once daily for 8 weeks
  Interventions: Dietary Supplement: omega 3 FA group
- VD3 and omega 3 FA group (Experimental): dietary supplement : VD3 and omega-3FA 50000 IU VD3/week for 8 weeks and 1000 mg wild salmon and fish oil complex (contain 300 mg of omega 3-FA) once daily for 8 weeks
  Interventions: Dietary Supplement: VD3 and omega- 3FA group
- control group (Experimental): no intervention was given
  Interventions: Other: control group

INTERVENTIONS:
Dietary Supplement: VD3 group — VD3 50000 IU/ week for 8 weeks
  Arms: VD3 group
Dietary Supplement: omega 3 FA group — omega 3 FA group 300 mg once daily for 8 weeks
  Arms: omega 3- FA group
Dietary Supplement: VD3 and omega- 3FA group — 50000 IU VD3/week for 8 weeks and 300 mg of omega- 3 FA once daily for 8 weeks
  Arms: VD3 and omega 3 FA group
Other: control group — no intervention was given
  Arms: control group

SUMMARY:
The Combined effect of Vitamin D3 and Omega-3 supplements on serum leptin and Glycated hemoglobin (Hb A1C) levels in Jordanian people with vitamin D deficiency.

DETAILED DESCRIPTION:
Nothing is published in the literature about effect of vitamin D3 (VD3) and omega-3 fatty acids (omega-3FA) on serum leptin and glycated hemoglobin ( HbA1C)

This study will be conducted to investigate effect of VD3 and omega-3FA alone and with each other on serum leptin and Glycated hemoglobin (Hb A1C) levels in Jordanian people with vitamin D deficiency.

This randomized, controlled clinical trial will be designed to test effects of 50,000 IU VD3 weekly and 1000 mg omega-3FA daily for eight weeks, separately and with each other, on on serum leptin and Glycated hemoglobin (Hb A1C) levels .

ELIGIBILITY:
Inclusion Criteria:

* jordanian people aged 25-55
* medical diagnosis of vitamin D deficiency ( VD <25 ng/ ml)

Exclusion Criteria:

* Blood disorders including
* thalassemia
* sickle cell disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
VD 3 | 8 weeks
  Serum level of 25-hydroxyvitamin D
leptin | 8 weeks
  serum level of leptin
HbA1C | 8 weeks
  plasma concentration of HbA1C

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Principal Investigator — Applied Science Private University
Locations (1):
- Applied Science University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underline results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: when summary data will published
Access Criteria: open access

REFERENCES:
- [Result] Ross AC. The 2011 report on dietary reference intakes for calcium and vitamin D. Public Health Nutr. 2011 May;14(5):938-9. doi: 10.1017/S1368980011000565. No abstract available. PMID 21492489